CLINICAL TRIAL: NCT06404281
Title: Anti-PD-1 Antibody Armored γδ T Cells in the Treatment of Advanced Solid Tumors, a Phase I Clinical Trail
Brief Title: γδ T-PD-1 Ab Cells in the Treatment of Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Changzhou No.2 People's Hospital (Other)
Responsible Party: Principal Investigator, Hua Jiang, Chief Director of Oncology Department, Changzhou No.2 People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: [2024]KY024-01
Record Dates: First submitted 2024-04-21; First posted 2024-05-08 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- γδ T-PD-1 Ab cells (Experimental): Patients will receive 6 cycles of ex-vivo expanded γδ T-PD-1 Ab cells treatments,at two-weeks' intervals.γδ T-PD-1 Ab cells are transfused to patients in atypical 3+3 dose-escalation design(Dose escalation,3x10^7/kg,1x10^8/kg,3x10^8/kg).
  Interventions: Biological: γδ T-PD-1 Ab cells

INTERVENTIONS:
Biological: γδ T-PD-1 Ab cells — Cells will be extracted from a healthy donor, followed by ex-vivo expansion, activation and genetic engineering. The ex-vivo expanded γδ T-PD-1 Ab cells will be adoptively transfused to tumor patients.

SUMMARY:
This study intends to combine the advantages of γδ T cells and PD-1 monoclonal antibody to conduct an exploratory clinical study on the safety and efficacy of PD-1 antibody armored γδ T cells (γδ T-PD-1 Ab cells) in the treatment of advanced solid tumors.

DETAILED DESCRIPTION:
This is a single-center, single-arm, phase I clinical trial to evaluate the safety and efficacy of γδ T-PD-1 Ab cells in patients with advanced solid tumors without standard treatment. A typical 3+3 dose-escalation design will be used to determine the optimal dose level of γδ T-PD-1 Ab cells based on the incidence of dose-limiting toxicity (DLT). The initial infusion dose level will start from 3×10^7/kg to 3×10^8/kg in every 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. The patient voluntarily signs the informed consent and can complete the follow-up examination, evaluation and treatment;
2. Age 18-80 years old, gender is not limited;
3. The histopathological diagnosis was malignant solid tumor;
4. Clinical or pathological was stage IV according to AJCC 8th edition stage;
5. Subjects with advanced solid tumors without standard treatment options;
6. ECOG score 0-1;
7. Expected survival ≥6 months;
8. Have at least one evaluable lesion according to RECIST 1.1 criteria;
9. Organ function level requirements (no blood transfusion or blood products, no hematopoietic stimulating factors, no albumin or blood products used within 14 days prior to the first dose);
10. Bone marrow function: absolute value of neutrophils (ANC) ≥1.5×109, platelets ≥75×109, and hemoglobin (Hb) ≥90g/L;
11. Liver function: total bilirubin ≤1.5 times the upper limit of normal (ULN); Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 times ULN (5.0 times ULN if liver metastasis is present), alkaline phosphatase < 5 × ULN;
12. Renal function: serum creatinine level ≤2 ULN, creatinine clearance > 50mL/min (according to Cockcroft-Gault formula); Urine protein <2+(If urine protein ≥2+, urine protein measurement should be collected for 24 hours, and the total amount should be <1g to be allowed to enter the group);
13. The serum pregnancy test of women of childbearing age in the 7 days prior to Gamma-delta T-PD-1 Ab infusion is negative, and any fertile male and female subject must consent to the use of an effective contraceptive method throughout the study and for at least 12 weeks after the last study administration. In the researchers' judgment, a subject is fertile: he/she is biologically capable of having children and having a normal sex life.
14. A hysterectomy or bilateral oophorectomy has been performed, or ovarian failure has been medically confirmed, or post-menopause has been medically confirmed (menopause for at least 12 consecutive months without pathological or physiological causes).

Exclusion Criteria:

1. Intolerance or allergy to any ingredient or similar drug in the treatment plan planned for this study;
2. Metastasis of symptomatic central system;
3. Have received other cell therapies, including NK, CIK, DC, CTL, CAR-T, TCR-T, and stem cell therapy in the past 4 weeks;
4. Received systemic steroid therapy (> 10 mg/kg prednisone or equivalent) or any other form of immunosuppressive medication within two weeks prior to the first dose; Corticosteroids (≤10mg oral prednisone or equivalent) were used in subjects with chronic obstructive pulmonary disease, saline corticosteroids (such as hydrohydrocortisone) were used in subjects with postural hypotension, and low-dose supplemental corticosteroids were used in subjects with adrenal insufficiency.
5. Plan to use any other form of systemic antitumor therapy during the study period;
6. History of known hematological malignancy, primary brain tumor or sarcoma, or other primary solid tumor within 6.5 years, unless cured and no evidence of recurrence of the disease within 5 years. With the exception of cured basal cell carcinoma of the skin and cervical carcinoma in situ;
7. History of interstitial lung disease, non-infectious pneumonia or uncontrolled disease, including pulmonary fibrosis and acute lung disease;
8. Active autoimmune diseases within the past 2 years requiring systemic treatment (such as glucocorticoids or immunosuppressive drugs), and related replacement therapy (such as thyroxine, insulin, or physiologic glucocorticoid replacement therapy for renal or pituitary insufficiency); Bisphosphonates were administered within 2 months prior to Γδ T-PD-1 Ab infusion.
9. Known subjects had systemic vasculitis, co-active or uncontrolled autoimmune disease, primary or secondary immune deficiency, graft-versus-host disease (GvHD).
10. Hepatitis B infection, hepatitis C infection, human immunodeficiency virus (HIV) infection, Treponema pallidum (TP) infection.
11. Had undergone major surgery within 4 weeks prior to screening that was assessed by the investigator as unsuitable for enrollment.
12. Acute infection and gastrointestinal bleeding occurred in 4 weeks.
13. Major organ dysfunction: absolute value of neutrophils (ANC) < 1.5×109, platelets < 75×109, and hemoglobin (Hb) < 90g/L; Serum albumin < 28g/L, total bilirubin >51μmol/L, alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >5 times the upper limit of normal, creatinine > 1.5 times the upper limit of normal; Have abnormal coagulation function (INR > 1.5 or PT >1.2 ULN or PTT >1.2 ULN), have a tendency to bleed, or are receiving thrombolytic or anticoagulant therapy.
14. The subject's heart meets any of the following conditions: Left ventricular ejection fraction (LVEF) ≤45%; New York Heart Association (NYHA) Class III or IV congestive heart failure; QTcB > 450 msec; Other heart conditions that the investigators judged unsuitable for inclusion.
15. People with a history of epilepsy or other active central nervous system diseases.
16. Received live vaccine within 6 weeks prior to screening, and received hematopoietic stimulating factors, such as colony-stimulating factor and erythropoietin, within 2 weeks prior to treatment; Major surgical procedures (excluding diagnostic surgical procedures) within 4 weeks before the start of treatment;
17. Evidence of uncontrolled and severe active infection at the time of screening (e.g., sepsis, bacteremia, fungemia), or a recent (within 4 months) history of deep tissue infection (e.g., fasciitis or osteomyelitis).
18. Participate in other interventional clinical investigators within 3 months prior to infusion of γδ T-PD-1 AB-PD-1 Ab.
19. A known mental or substance abuse disorder may interfere with the requirement to cooperate in the completion of the trial.
20. Women who are pregnant or breastfeeding, or who plan to become pregnant or have children during the study period.
21. In the investigator's judgment, the subject has any serious acute or chronic physical or mental illness, or laboratory abnormalities that could increase the risk of study participation, study administration, or possibly affect the interpretation of study results.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Safety evaluation: Incidence of Adverse events (AEs) | up to 60 weeks
  Therapy-related adverse events will be recorded and assessed according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE, Version 5.0).
Safety evaluation: Dose limited toxicity (DLTs) | up to 60 weeks
  The incidence, characteristic and severity of DLTs will be recorded and assessed.
Safety evaluation: Maximum-tolerated dose (MTD) | up to 60 weeks
  MTD or clinical recommended dose will be recorded and evaluated.

SECONDARY OUTCOMES:
Efficacy evaluation: Objective Response Rate(ORR) | up to 15months
  Objective response rate will be assessed by investigators.
Efficacy evaluation: Disease Control Rate (DCR) | up to 15months
  Disease Control Rate will be assessed by investigators.
Efficacy evaluation: Progress Free Survival(PFS) | up to 15months
  Observation for progression-free survival (PFS) will be recorded until 15 months after the start of 1st cycle of treatment.
Efficacy evaluation: Overall Survival (OS) | up to 15months
  Observation for overall survival (OS) will be recorded until 15 months after the start of 1st cycle of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Hua Jiang, MD, Study Director — Changzhou No.2 People's Hospital
Locations (1):
- Changzhou No.2, Changzhou, China

IPD SHARING:
Plan to Share IPD: No